CLINICAL TRIAL: NCT05271708
Title: Explore the Short- and Mid-term Effects of Fespixon in Scar Cosmesis Following Cervical or Abdominal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Shao-Cheng Liu, Associate Professor, National Defense Medical Center, Taiwan
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B202105176; B202105176L (Other: Tri-Service General Hospital, National Defense Medical Center)
Record Dates: First submitted 2022-02-15; First posted 2022-03-09 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Scar
Keywords: Fespixon; Thyroidectomy; caesarean section; Scar; ON101
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Intervention Model Description: The patient's wound was treated with a placebo or therapeutic ointment on the right side and a placebo or therapeutic ointmenton the left side.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcomes (VSS score) assessors do not know which side is applied with the therapeutic ointment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fespixon cream (Experimental): Fespixon cream contains 1.25% extracts of Plectranthus amboinicus (PA-F4, 0.25%) and Centella asiatica (S1, 1%) with appearance in yellow-green to light green color. Fespixon cream will be applied twice daily for up to 12 weeks to the linear wound.
  Interventions: Drug: Fespixon cream
- Placebo Cream (Placebo Comparator): Placebo cream with appearance in yellow-green to light green color, same appearance as Fespixon cream, will be applied twice daily for up to 12 weeks to the linear wound.
  Interventions: Drug: Placebo Cream

INTERVENTIONS:
Drug: Fespixon cream — Bounded by the midpoint of the scar, each patient received two topical scar formulations consisting of Fespixon cream on one side, and placebo cream on the other side. Treatment was given twice a day for 84 days.
  Other Names: ON101 cream
  Arms: Fespixon cream
Drug: Placebo Cream — Bounded by the midpoint of the scar, each patient received two topical scar formulations consisting of Fespixon cream on one side, and placebo cream on the other side. Treatment was given twice a day for 84 days.
  Arms: Placebo Cream

SUMMARY:
The aim of this study is to evaluate the efficacy of the Fespixon cream for prevention and/or appearance reduction of different types of linear scars during the 12-week treatment phase, which is assessed by the blinded independent evaluator.

DETAILED DESCRIPTION:
Methods: This study was designed as a prospective, double-blind, placebo-controlled trial involving 50 patients with linear scars. Bounded by the midpoint of the scar, each patient received a topical scar formulation consisting of fespixon cream on one side of scar, and placebo cream on the other side of scar. Treatment was given twice a day for 84 days. Assessments of the scars were performed at visit 1, 2, 3 following the onset of topical application using three methods: a clinical assessment using the Vancouver Scar Scale/ modified Vancouver Scar Scale, a photographic assessment to establish before and after treatment improvements, and at the end of the study period, patients completed a final satisfaction questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged over 20 years old (inclusive).
2. Subjects with linear scar in neck or abdomen following elective surgery, including thyroid and parathyroid surgery, excision of neck mass, caesarean section, trans-abdominal hysterectomy, trans-abdominal myomectomy or any neck or abdominal surgeries which can be managed by primary closure of clean surgical wounds.

Exclusion Criteria:

1. Subjects who have previous neck or abdominal trauma that will affect the surgical incision site.
2. After radiation therapy for cervical/abdominal cancer, or previous medical history with chemo-therapy or targeted therapy for any reason.
3. Laboratory values at Screening of:

   Note: The investigator will decide which of the following laboratory tests should be performed considering the condition of the subject.
   1. Albumin < 2.5 g/dL (for subjects with severe malnutrition)
   2. HbA1c >12.0% (for subjects with severe diabetes)
   3. Liver function test [ aspartate aminotransferase (AST) and alanine transaminase (ALT)] > 3x the upper limit of normal
   4. Renal function test [Serum Creatinine] > 2x the upper limit of normal
4. Subject is currently receiving immunosuppressant or systemic corticosteroids.
5. Has any other factor which may, in the opinion of the investigator, compromise participation in the study.(Including subjects with medical history of keloid or hypertrophic scar).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
VSS total scores at Day 1 and Week 12 assessed by 3 blind evaluators | 12-week
  The VSS scores, assessed by 3 blind evaluators, changed from Day 1 to Week 12 will be used as an objective evidence.

SECONDARY OUTCOMES:
mVSS individual scores at Day 1 and Week 12 assessed by a Principal Investigator | 12-week
  The mVSS scores, assessed by a Principal Investigator, changed from Day 1 to Week 12 will be used as an auxiliary evidence.
Hue feature-Red values via digital analysis at Day 1 and Week 12 | 12-week
  1. Using the data of Day1 as baseline, relative Δ ratio represents the difference of Δ ratio between Week 12 and Day1 out of baseline.
  NOTE1: Relative Δ ratio = (Week 12 Δ ratio - Day1 Δ ratio)/ Day1 Δ ratio
  NOTE2: Difference ratio= Δ ratio = Δ(scar-skin)/skin
Hue feature-Green values via digital analysis at Day 1 and Week 12 | 12-week
  1. Using the data of Day1 as baseline, relative Δ ratio represents the difference of Δ ratio between Week 12 and Day1 out of baseline.
  NOTE1: Relative Δ ratio = (Week 12 Δ ratio - Day1 Δ ratio)/ Day1 Δ ratio
  NOTE2: Difference ratio= Δ ratio = Δ(scar-skin)/skin
Hue feature-Blue values via digital analysis at Day 1 and Week 12 | 12-week
  1. Using the data of Day1 as baseline, relative Δ ratio represents the difference of Δ ratio between Week 12 and Day1 out of baseline.
  NOTE1: Relative Δ ratio = (Week 12 Δ ratio - Day1 Δ ratio)/ Day1 Δ ratio
  NOTE2: Difference ratio= Δ ratio = Δ(scar-skin)/skin
CIELab-lightness values via digital analysis at Day 1 and Week 12 | 12-week
  1. Using the data of Day1 as baseline, relative Δ ratio represents the difference of Δ ratio between Week 12 and Day1 out of baseline.
  NOTE1: Relative Δ ratio = (Week 12 Δ ratio - Day1 Δ ratio)/ Day1 Δ ratio
  NOTE2: Difference ratio= Δ ratio = Δ(scar-skin)/skin
CIELab-a values via digital analysis at Day 1 and Week 12 | 12-week
  1. Using the data of Day1 as baseline, relative Δ ratio represents the difference of Δ ratio between Week 12 and Day1 out of baseline.
  NOTE1: Relative Δ ratio = (Week 12 Δ ratio - Day1 Δ ratio)/ Day1 Δ ratio
  NOTE2: Difference ratio= Δ ratio = Δ(scar-skin)/skin
CIELab-b values via digital analysis at Day 1 and Week 12 | 12-week
  1. Using the data of Day1 as baseline, relative Δ ratio represents the difference of Δ ratio between Week 12 and Day1 out of baseline.
  NOTE1: Relative Δ ratio = (Week 12 Δ ratio - Day1 Δ ratio)/ Day1 Δ ratio
  NOTE2: Difference ratio= Δ ratio = Δ(scar-skin)/skin
Textual features-Contrast (Con) values via digital analysis at Day 1 and Week 12 | 12-week
  1. Using the data of Day1 as baseline, relative Δ ratio represents the difference of Δ ratio between Week 12 and Day1 out of baseline.
  NOTE1: Relative Δ ratio = (Week 12 Δ ratio - Day1 Δ ratio)/ Day1 Δ ratio
  NOTE2: Difference ratio= Δ ratio = Δ(scar-skin)/skin
Textual features-Homogeneity (Hom) values via digital analysis at Day 1 and Week 12 | 12-week
  1. Using the data of Day1 as baseline, relative Δ ratio represents the difference of Δ ratio between Week 12 and Day1 out of baseline.
  NOTE1: Relative Δ ratio = (Week 12 Δ ratio - Day1 Δ ratio)/ Day1 Δ ratio
  NOTE2: Difference ratio= Δ ratio = Δ(scar-skin)/skin
Textual features-Correlation (Cor) values via digital analysis at Day 1 and Week 12 | 12-week
  1. Using the data of Day1 as baseline, relative Δ ratio represents the difference of Δ ratio between Week 12 and Day1 out of baseline.
  NOTE1: Relative Δ ratio = (Week 12 Δ ratio - Day1 Δ ratio)/ Day1 Δ ratio
  NOTE2: Difference ratio= Δ ratio = Δ(scar-skin)/skin
Textual features-Entropy (ENT) values via digital analysis at Day 1 and Week 12 | 12-week
  1. Using the data of Day1 as baseline, relative Δ ratio represents the difference of Δ ratio between Week 12 and Day1 out of baseline.
  NOTE1: Relative Δ ratio = (Week 12 Δ ratio - Day1 Δ ratio)/ Day1 Δ ratio
  NOTE2: Difference ratio= Δ ratio = Δ(scar-skin)/skin
VAS (Visual Analogue Scale) score at Week 12 | 12-week
  VAS score (on a scale from 0 to 10) at Week 12 are used to present the satisfaction of participants. Zero means participants feel "not at all satisfied" and 10 means participants feel "completely satisfied".

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Cheng Liu, PhD, Principal Investigator — Tri-Service General Hospital, National Defense Medical Center
Locations (1):
- Tri-Service General Hospital, National Defense Medical Center, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No